CLINICAL TRIAL: NCT06908928
Title: An Open-Label, Multicenter, Phase Ib Dose Randomization Study of Bulumtatug Furvedotin (BFv; 9MW2821) in Subjects With Recurrent or Metastatic Triple-Negative Breast Cancer Previously Treated With Antibody-Drug Conjugates
Brief Title: A Dose Randomization Study of Bulumtatug Fuvedotin in TNBC Patients Previously Treated With ADCs
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-2022-CP103
Record Dates: First submitted 2025-03-20; First posted 2025-04-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Cancer
Keywords: 9MW2821; bulumtatug fuvedotin
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose level 1 of BFv (Experimental)
  Interventions: Drug: bulumtatug fuvedotin
- Dose level 2 of BFv (Experimental)
  Interventions: Drug: bulumtatug fuvedotin

INTERVENTIONS:
Drug: bulumtatug fuvedotin — given via intravenous infusion on day 1 and day 8 of every 21-day cycle at dose level 1
  Arms: Dose level 1 of BFv
Drug: bulumtatug fuvedotin — given via intravenous infusion on day 1 and day 8 of every 21-day cycle at dose level 2
  Arms: Dose level 2 of BFv

SUMMARY:
The goal of this clinical trial is to investigate if treatment with bulumtatug fuvedotin is effective in triple-negative breast cancer patients who have previously received treatment with an antibody-drug conjugates.

ELIGIBILITY:
Inclusion Criteria

* Patient has measurable disease by RECIST v1.1
* Recurrent or metastatic triple-negative breast cancer patients as per current ASCO/CAP guidelines
* Patient has received prior treatment with a taxane and an antibody-drug conjugate with a topoisomerase inhibitor payload.
* Patient has received no more than 3 prior lines of cytotoxic therapy in the locally advanced or metastatic setting.
* Provision of archival tumor tissue or fresh tumor biopsy.
* Capable of giving informed consent
* Male or female subjects aged ≥ 18 years.
* Subjects must be willing to receive blood transfusions if medically indicated.
* ECOG 0-1
* Adequate hematologic and organ function
* Life expectancy of at least 3 months as assessed by the investigator
* Compliance with contraceptive requirement

Exclusion Criteria:

* Have received any prior treatment with enfortumab vedotin, tisotumab vedotin or other MMAE based or nectin-4 targeted antibody-drug conjugates.
* Unstable CNS metastasis requiring treatment in the last 28 days.
* Acute infection requiring IV treatment in the last 14 days.
* Grade ≥2 peripheral neuropathy.
* Pregnant or breastfeeding women.
* Life-threatening illness or uncontrolled medical conditions that could compromise the subject's safety or put the study outcomes at risk
* Any systemic anticancer therapy in the last 28 days prior to first administration of study drug.
* Active HCV, HBV or HIV infection unless well controlled with anti-viral therapy.
* Active or chronic corneal disorder, keratitis, corneal ulcerations or Sjogren's syndrome.
* Have any ongoing acute inflammatory skin disease or chronic skin disease not well controlled.
* Have been diagnosed with another primary malignancy except for adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or subjects with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
* Have significant, uncontrolled or active cardiovascular disease
* Have active or a history of pneumonitis or interstitial lung disease that requires corticosteroid treatment. Patients with radiation pneumonitis that does not require treatment is allowed.
* Have uncontrolled diabetes.
* Have received any strong CYP3A4 inhibitors within 14 days prior to the first dose of study drug.
* Subjects known to be hypersensitive to bulumtatug fuvedotin or to any components of the formulation.
* History of drug abuse including narcotic and psychiatric drugs within 12 months prior to screening.
* Have received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to approximately 2 years
  Objective Response Rate according to RECIST v1.1 by investigator assessment

SECONDARY OUTCOMES:
Disease control rate | Up to approximately 2 years
  The percentage of patients who achieve complete response (CR), partial response (PR), or stable disease (SD) as per RECIST v1.1.
Clinical benefit rate | Up to approximately 2 years
  The percentage of patients who achieve CR, PR, or SD for at least 6 months.
Duration of response | Up to approximately 2 years
  The time from first documented response (CR or PR) to disease progression or death, whichever occurs first.
Progression-free survival | Up to approximately 2 years
  The time from treatment initiation to disease progression or death from any cause.
Overall survival | Up to approximately 2 years
  The time from treatment initiation to death from any cause.
Time to Maximum Concentration (Tmax) | Up to approximately 2 years
  Time to reach the maximum observed concentration of bulumtatug fuvedotin, TAb, and MMAE in blood.
Maximum Concentration (Cmax) | Up to approximately 2 years
  Maximum observed blood concentration of bulumtatug fuvedotin, TAb, and MMAE.
Half-life (t1/2) | Up to approximately 2 years
  The time required for the blood concentration of bulumtatug fuvedotin, TAb, and MMAE to decrease by 50%.
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Measurable Concentration (AUC0-t) | Up to approximately 2 years
  The area under the plasma concentration-time curve from time zero to the last measurable concentration for bulumtatug fuvedotin, TAb, and MMAE.
Incidence, rate and severity of treatment-emergent adverse events. | Up to approximately 2 years
  Incidence, rate and severity of AE, SAE, TRAE and AESI. Frequency of clinically significant abnormalities in physical examination, safety laboratory tests, urinalysis, vital signs, and 12-Lead ECG record. Safety will be reported as incidence and rate of treatment-emergent adverse events using NCI CTCAE v5.0 criteria.
Immunogenicity | Up to approximately 2 years
  Incidence and rates of ADA and Nab.
Immunogenicity | Up to approximately 2 years
  Titre of ADA and Nab.

OTHER OUTCOMES:
Efficacy parameters and biomarkers including but not limited to nectin-4 expression level. | Up to approximately 2 years
  The proportion of nectin-4 positive and negative patients. The proportion of nectin-4 positive patients who experienced objective response. The proportion of nectin-4 negative patients who experienced objective response.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - UChicago Medicine Comprehensive Cancer Center, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No